CLINICAL TRIAL: NCT02021045
Title: Quantity, Quality and Laterality of Cerebral Microembolism During Veno-Venous Hemodialysis.
Brief Title: Cerebral Microembolism During Hemodialysis
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Gabor Erdoes, Dr Gabor Erdoes, Medical University of Vienna
Other Study IDs: 1706/2013
Record Dates: First submitted 2013-11-20; First posted 2013-12-27 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Complication of Dialysis; Thrombus Due to Renal Dialysis Device, Implant, or Graft; Cerebral Embolism
MeSH Terms: conditions — Intracranial Embolism | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient on Hemodialysis: Renal hemodialysis
  Interventions: Device: Renal hemodialysis (Fresenius 2008K, Bad Homburg, Germany)
- Patient in a hemodialysis-free interval: No Renal hemodialysis

INTERVENTIONS:
Device: Renal hemodialysis (Fresenius 2008K, Bad Homburg, Germany) — Renal replacement therapy is frequently used in patients with renal failure in order to eliminate substances obligatory excreted by the urine.
  Other Names: Continuous veno-venous hemodialysis
  Groups: Patient on Hemodialysis

SUMMARY:
There is increasing evidence that renal replacement therapy (= continuous veno-venous hemodialysis) generates cerebral microembolism which is detectable on transcranial Doppler ultrasound.

The aim of this study is to monitor patients with transcranial Doppler under two conditions: during hemodialysis and in a hemodialysis-free interval (in each period cerebral embolic load is detected during 30 minutes).

The study hypothesis is that during hemodialysis the cerebral embolic load is significantly higher than in the hemodialysis-free interval.

ELIGIBILITY:
Inclusion Criteria:

* Renal replacement therapy (continuous veno-venous hemodilalysis) on the in-house intensive care unit
* Age > 18yrs and < 90yrs

Exclusion Criteria:

* Absent informed consent
* Preexistent neurological morbidity
* Neurocognitive disturbances
* Carotid artery stenosis > 70%
* Patent foramen ovale
* Treatment with other extracorporeal devices
* Cardial pathology (valvular heart disease, prosthesis, endocarditis)
* Pregnancy, drug abuse
* Inclusion in an other clinical study
* Allergy against materials of the medical device used in the study (transcranial Doppler) or temporal skin/bone lesions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population incloses patients who are in renal failure needing renal replacement therapy under intensive care conditions.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Quantity of cerebral embolic load | 30 minutes
  Cerebral embolic load is measured in a 30 minutes-interval during hemodialysis and in a hemodialysis-free interval.

SECONDARY OUTCOMES:
Quality and laterality of cerebral embolic load | 30 minutes
  Quality (solid vs. gaseous) and laterality (left vs. right hemispheric dominance) of cerebral embolic load is measured in a 30 minutes-interval during hemodialysis and in a hemodialysis-free interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria